CLINICAL TRIAL: NCT07134023
Title: Programme EducaTif d'Accompagnement pLuridisciplinaire Des Patientes Atteintes d'Endométriose
Brief Title: Educational Program for the Multidisciplinary Support of Patients With Endometriosis
Acronym: PETALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH2_DEFOUS_PETALE; ID RCB (Other: 2025-A00662-47)
Record Dates: First submitted 2025-08-07; First posted 2025-08-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: Endometriosis; Quality of life; Multidisciplinary; Nurse follow-up
MeSH Terms: conditions — Endometriosis | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group will participate in a therapeutic education and nursing support (Experimental): Therapeutic Education and Nursing Support Program for Supportive Care. In addition to conventional gynecological follow-up care, patients will participate in an initial educational assessment day. During this day, the patient will have a discussion with the pivot nurse to define personalized objectives, which will guide the choice of workshops and supportive care in the outpatient educational program.
  Interventions: Other: Supportive Care
- Control group (No Intervention): Patients follow conventional care.

INTERVENTIONS:
Other: Supportive Care — Initial Educational Assessment In addition to standard care, patients will meet the coordinating nurse for an initial educational assessment to evaluate their needs and present the multidisciplinary workshop program and individual support options. The nurse will register the patient for the first session, provide program materials, schedule the first follow-up call (1 month post-inclusion), and collect study questionnaires and demographics. If needed, the assessment may be scheduled within 15 days of inclusion.
  Educational Workshops Patients may attend workshops on topics like endometriosis, diet, sexuality, pain, fatigue, emotions, Pilates, non-drug symptom management, hypnoanalgesia, and fertility. At least three workshops are required, offered over two days.
  Telephone Follow-up Monthly calls for 6 months, then at 9 and 12 months, will monitor symptoms and refer patients to support services as needed.
  Arms: The experimental group will participate in a therapeutic education and nursing support

SUMMARY:
Background:

Endometriosis is a chronic gynecological condition characterized by the ectopic presence of endometrial tissue outside the uterine cavity. It affects approximately 2 to 10% of women of reproductive age and up to 50% of women with chronic pelvic pain. In France, between 1.5 and 2.5 million women are estimated to be affected. Endometriosis significantly impairs quality of life, with consequences on cognitive, behavioral, sexual, and emotional well-being, and has substantial socio-economic impact.

Rationale:

Current medical and surgical treatments primarily aim to reduce pain and preserve fertility but show limited effectiveness and are often discontinued due to adverse effects. Many women resort to self-management strategies, which may pose risks if not properly supervised. A multidisciplinary and integrative approach is essential to address the complex and multifactorial symptoms of endometriosis. Therapeutic patient education (TPE) is a recommended strategy that can empower patients in the management of chronic conditions, yet remains underdeveloped in endometriosis care pathways.

Objective:

This study aims to evaluate the effectiveness of a multidisciplinary educational program combined with nurse-led telephone follow-up on the quality of life of patients with endometriosis.

Methods:

The intervention will consist of a series of workshops led by various healthcare professionals (medical and paramedical), alongside regular nurse-led telephone follow-up. This approach intends to provide continuous support, assess patients' evolving needs, and facilitate access to supportive care services, particularly within regional endometriosis networks (ENDAURA and ENDOSUD).

Expected Outcomes:

The study will assess whether this intervention improves quality of life among women with endometriosis. It also aims to provide evidence for the scalability and transferability of such a program at a national level, in alignment with current public health priorities.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Age ≥ 18 years,
* Patient diagnosed with endometriosis confirmed by pelvic ultrasound and/or MRI,
* Patient experiencing chronic pelvic-perineal pain (± dysmenorrhea, dyspareunia, etc.) for at least 3 months,
* Ability to read and understand French,
* Affiliation with a social security system or equivalent.

Exclusion Criteria:

* Patient having already participated in an educational program or received multidisciplinary follow-up (involving at least 3 different healthcare professionals simultaneously within the same facility) in the past 12 months,
* Patient in an emergency situation, or under legal protection measures (guardianship, curatorship, or judicial protection) and unable to give consent,
* For patients at the experimental center only: inability to comply with study follow-up due to geographical, social, or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Endometriosis Health Profile-30 (EHP-30) | baseline (T0) to 6 months and 12 months (M12)
  Change in quality of life, measured by the Endometriosis Health Profile-30 (EHP-30) score, from baseline (T0) to 12 months (M12), in the experimental group receiving a multidisciplinary educational program with nurse-led telephone follow-up compared with the control group receiving standard care.

SECONDARY OUTCOMES:
Anxiety | baseline (T0), 6 months (M6), and 12 months (M12).
  Change in anxiety and depression scores, measured using the validated self-administered Hospital Anxiety and Depression Scale (HADS), between the experimental group and the control group at baseline (T0), 6 months (M6), and 12 months (M12).
  This 14-item questionnaire, rated from 0 to 3, is used to detect anxiety or depression. The score obtained for each component (seven items for the anxiety component and seven items for the depression component) is analyzed. The maximum possible score for each component is 21. A score of seven or less indicates an absence of symptoms; a score between eight and 10 indicates possible symptoms; and a score of 11 or more indicates definite symptoms.
Score of the the brief pain inventory | baseline (T0), 6 months (M6), and 12 months (M12).
  Change in pain scores, assessed using the Brief Pain Inventory (BPI), a validated self-administered questionnaire evaluating pain location, intensity, and interference with daily activities, between the experimental group and the control group at baseline (T0), 6 months (M6), and 12 months (M12).
  This self-questionnaire allows you to evaluate various aspects of pain, such as its location, intensity, and frequency. Pain intensity is evaluated using a scale from 0 to 10, where 0 indicates no pain and 10 indicates the most severe pain imaginable.
dyspareunia and dysmenorrhea | baseline (T0), 6 months (M6), and 12 months (M12)
  Change in pain scores related to dyspareunia and dysmenorrhea, assessed using a Visual Analogue Scale (VAS), between the experimental group and the control group at baseline (T0), 6 months (M6), and 12 months (M12).
  This validated self-administered scale allows participants to rate the intensity of their pain along a continuous line, typically 0-10, where higher scores indicate greater pain.
Female Sexual Function | baseline (T0), 6 months (M6), and 12 months (M12).
  Change in sexual function, assessed using the Female Sexual Function Index (FSFI), a validated self-administered questionnaire evaluating sexual function in women, between the experimental group and the control group at baseline (T0), 6 months (M6), and 12 months (M12).
  This self-report questionnaire assesses sexual function in women. It contains 19 items, which are divided into six domains. Each item is rated on a scale from 0 to 6. The total score is obtained by adding together the scores for each domain. Higher scores indicate better sexual function and quality of life.
Sleep | baseline (T0), 6 months (M6), and 12 months (M12).
  Change in sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-administered questionnaire evaluating sleep disturbances and overall sleep quality, between the experimental group and the control group at baseline (T0), 6 months (M6), and 12 months (M12).
  PSQI is a validated, 19-item, self-administered questionnaire that measures sleep problems. A score of 5 or less indicates "good sleepers," while a score strictly greater than 5 indicates "poor sleepers."
Hormonal treatments | baseline (T0) to 12 months
  Use of hormonal treatments, including information on the International Nonproprietary Name (INN), daily dosage, and duration of use, in the experimental group versus the control group from baseline (T0) to 12 months (M12)
Analgesic medications | baseline (T0) to 12 months
  Use of analgesic medications, including the INN, daily dosage, and duration of use, in the experimental group versus the control group from baseline (T0) to 12 months (M12).
medical consultations, hospitalizations, and work absences | baseline (T0) to 12 months (M12)
  Number of medical consultations, hospitalizations, and work absences related to endometriosis between the experimental group and the control group from baseline (T0) to 12 months (M12).
the type and frequency of supportive care interventions | baseline (T0) and 12 months (M12)
  Type and frequency of supportive care interventions used by patients in the experimental group versus the control group between baseline (T0) and 12 months (M12).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Axium, Aix-en-Provence
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay

IPD SHARING:
Plan to Share IPD: No
The study sponsor is the owner of the data and no use or transmission to a third party may be made without its prior consent. All information resulting from this clinical research protocol is considered confidential.